CLINICAL TRIAL: NCT04847765
Title: A Pilot Study to Assess the Procedural Feasibility to Combine and Compare Dynamic Magnetic Resonance Imaging and an Isovolumetric Intragastric Balloon to Assess Gastric Contractility in Healthy Adults
Brief Title: ANTERO-6 Cine-MRI Study
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Universitaire Ziekenhuizen KU Leuven (Other)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Device Feasibility
Other Study IDs: S65104
Record Dates: First submitted 2021-04-09; First posted 2021-04-19 (Actual); Last update posted 2021-09-30 (Actual); Status verified 2021-09

CONDITIONS: Health

STUDY DESIGN:
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (1):
- Combined pressure measurement and MRI (Experimental): Gastric motility is evaluated simultaneously by means of the investigational medical device and by means of cine-MRI.
  Interventions: Device: VIPUN Gastric Monitoring System prototype

INTERVENTIONS:
Device: VIPUN Gastric Monitoring System prototype — The VIPUN Balloon Catheter prototype is a nasogastric feeding tube with integrated balloon that can be inflated with a preset volume of air. Intraballoon pressure changes are recorded outside the body. Gastric contractions can be detected in the pressure profile.
  The recording lasts 30 minutes and is combined with simultaneous cine magnetic resonance imaging.

SUMMARY:
Previous research by TARGID (KU Leuven) has demonstrated the feasibility to assess gastric content volume by means of magnetic resonance imaging (MRI) while simultaneously evaluating gastric motor function by means of an isovolumetric balloon technique. This and other research concluded that in general, the motility readout of the isovolumetric balloon is associated with gastric contractions.

However, the exact relation between individual gastric contractions and individual intraballoon pressure waves remains incompletely understood.

Simultaneous assessment of gastric motility by means of an isovolumetric balloon and dynamic cine-MRI can validate that slow, high-amplitude intraballoon pressure waves are indeed induced by gastric muscle contractions. This evaluation might also enable us to attribute artefacts present in the pressure signal to physiologic processes such as cardiac, respiratory, intestinal and whole-body movements.

To date substantial uncertainty exists on the optimal procedural approach to evaluate gastric motility simultaneously with cine-MRI and the isovolumetric balloon.

The aim of this pilot study is to verify the feasibility of a several aspects of a larger confirmatory study protocol. This includes the evaluation of contrast of the balloon catheter on MRI (this would omit the need for radiographic confirmation), timelines, practical hurdles, analysis procedures and data management.

ELIGIBILITY:
Inclusion Criteria:

* Signed Informed Consent
* At least 18 years old
* Male
* BMI between and including 18 and 30
* Understand and able to read Dutch
* In good health on the basis of medical history

Exclusion Criteria:

* Using any medication that might affect gastric function or visceral sensitivity
* Known / suspected current use of illicit drugs
* Known psychiatric or neurological illness
* Any gastrointestinal surgery that could influence normal gastric function in the opinion of the Investigator
* History of heart or vascular diseases like irregular heartbeats, angina or heart attack
* Nasopharyngeal surgery in the last 30 days
* History of thermal or chemical injury to upper respiratory tract or esophagus
* Current esophageal or nasopharyngeal obstruction
* Known coagulopathy
* Known esophageal varices
* Metal or other MRI incompatible implants
* Contra-indications for MR (checked by MR safety questionnaire)
* Claustrophobia

Min Age: 18 Years | Sex: Male | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 2 (Actual)
Dates: Start 2021-04-21 (Actual); Primary Completion 2021-04-30 (Actual); Study Completion 2021-04-30 (Actual)

PRIMARY OUTCOMES:
Time of gastric contractions identified by means of the investigational medical device | 30 minutes
  Analysis software filters the pressure signal and identifies individual gastric contractions.
  The exact time at which each contraction is detected within a 30-minute recording period is documented.
Gastric contractions identified visually by an expert radiologist | 30 minutes
  The exact time at which each gastric contractile event is most clearly visible within a 30-minute recording period is documented.

CONTACTS AND LOCATIONS:
Locations (1):
- UZ Leuven, Leuven, Belgium